CLINICAL TRIAL: NCT03653455
Title: Patient Outcomes Collection: How Can we do Better? A Randomized Trial to Determine Factors Which May Affect Patient Compliance.
Brief Title: Patient Outcomes Collection: How Can we do Better?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: American Orthopaedic Society for Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18041709
Record Dates: First submitted 2018-07-24; First posted 2018-08-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
Keywords: Shoulder; Arthroscopy; sub-acromial decompression; distal clavicle resection; biceps tenodesis; rotator cuff repair; Patient reported outcomes
MeSH Terms: conditions — Shoulder Pain | interventions — Lead

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre- and post-operative discussion group (Experimental): Patients will discuss with their care provider their health outcomes before and at 6-months after their surgery. In addition, patients will receive email reminders to complete their forms, if they haven't done so.
  Interventions: Behavioral: Email reminders; Behavioral: Pre- and Post-operative discussion
- Incentivised group (Experimental): Patients will receive up to $30 in amazon gift cards as an incentive if they complete their forms before surgery, as well as at 6-months and 1-year after surgery. In addition, patients will receive email reminders to complete their forms, if they haven't done so.
  Interventions: Behavioral: Email reminders; Behavioral: Incentive
- Control group (Experimental): Patients will only receive email reminders to complete their forms, if they haven't done so.
  Interventions: Behavioral: Email reminders

INTERVENTIONS:
Behavioral: Email reminders — Patients will receive email reminders until their PROs are completed.
Behavioral: Pre- and Post-operative discussion — Patients will discuss with their provider the importance of PROs pre-operatively, as well as their post-operative progression in comparison to established norms.
  Arms: Pre- and post-operative discussion group
Behavioral: Incentive — Patients will receive up to $30 in amazon gift cards upon the completion of their PROs.
  Arms: Incentivised group

SUMMARY:
Patient reported outcomes (PROs) are widely used by clinical providers as important tools to help inform their clinical and research practice, and to improve quality of care for patients. In this study, the investigators aim to investigate ways by which patient PRO completion rates may be improved.

DETAILED DESCRIPTION:
Patient reported outcomes (PROs) are widely used by clinical providers as important tools to help inform their clinical and research practice, and to improve quality of care for patients. In addition, PROs are increasingly cited as a tool in measuring surgical performance and the value of health care services being delivered. The quality of data captured by PROs is, however, largely dependent on patients' response rates, both pre- and post-operatively. For pre-operative surveys, higher response rates may be achieved as patients may be reminded to complete their surveys at an office visit or prior to surgery. However, patient non-compliance presents a major challenge post-operatively, undermining PRO data integrity.

As clinical practices have moved to using PROs for all patients, rather than just a research tool, automated systems have been developed to deliver and collect PRO electronically. However, while automation has helped streamline PRO administration and data collection, this hasn't always translated into obtaining better PRO compliance rates. In an attempt to improve response rates, efforts have been made to reduce patient burden (by reducing the number of questions asked, for example), to regularly remind patients to complete their forms (either by email or telephone), or even offer patients monetary or non-monetary incentives.

Despite these measures' variable success, however, achieving high response rates remains a challenge. This, in part, is due to the fact these platforms depend heavily on patients receiving the request and their willingness to participate in the program, often long after their care is completed. As data are increasingly used to measure physician performance and quality, as well as to determine reimbursement, low patient compliance rates remain a significant impediment and affect the validity of the data.

In this study, the invetigators hypothesize that direct patient engagement can improve patient compliance with automated PRO capture.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo shoulder arthroscopy for rotator cuff condition (sub-acromial decompression, distal clavicle resection, biceps tenodesis, partial or full thickness rotator cuff tear repair or debridement) will be eligible for enrollment in the appropriate cohort. There will be no restrictions to this enrollment apart from that presented in the exclusions below.

Exclusion Criteria:

1. Minors or those over the age of 80
2. Subjects lacking English proficiency to complete the PROs of interest.
3. Past or current medical history that would preclude patients from undergoing surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Does patient engagement, through education or monetary incentivization, increase PRO compliance rate at 1 year after surgery, when compared to PRO compliance rate before surgery? | Change in PRO compliance rate between pre-surgery and 1-year post surgery
  Patients will discuss the importance of PROs and how they can be used to predict their health outcome with their care provider. Alternatively, patients may receive amazon gift cards if they complete their PROs before surgery, as well as at 6-months and 1-yr after surgery. Three established PROs [American Shoulder And Elbow Surgeons (ASES), Single Assessment Numeric Evaluation (SANE), and the Veteran Rand 12-Item and 12-Item Short Form Health Survey (VR/SF12)] will be automatically emailed to patients using an electronic platform (OBERD). Rate at which these forms are completed (compliance rate) before surgery, as well 1-year post surgery will be monitored through OBERD.

SECONDARY OUTCOMES:
Effects of age on PRO compliance rate. | Change in PRO compliance rate between pre-surgery and 1-year post surgery
  Assess how patients' age might change PRO compliance from baseline (before surgery) to 1-year after surgery. Three established PROs [American Shoulder And Elbow Surgeons (ASES), Single Assessment Numeric Evaluation (SANE), and the Veteran Rand 12-Item and 12-Item Short Form Health Survey (VR/SF12)] will be automatically emailed to patients using an electronic platform (OBERD). Rate at which these forms are completed (compliance rate) before surgery, as well 1-year post surgery will be monitored through OBERD.
Effects of technological literacy on PRO compliance rate. | Change in PRO compliance rate between pre-surgery and 1-year post surgery
  Assess how technological literacy might change PRO compliance from baseline (before surgery) to 1-year after surgery. Three established PROs [American Shoulder And Elbow Surgeons (ASES), Single Assessment Numeric Evaluation (SANE), and the Veteran Rand 12-Item and 12-Item Short Form Health Survey (VR/SF12)] will be automatically emailed to patients using an electronic platform (OBERD). Rate at which these forms are completed (compliance rate) before surgery, as well 1-year post surgery will be monitored through OBERD.
Effects of English proficiency on PRO compliance rate. | Change in PRO compliance rate between pre-surgery and 1-year post surgery
  Assess how English proficiency might change PRO compliance from baseline (before surgery) to 1-year after surgery. Three established PROs [American Shoulder And Elbow Surgeons (ASES), Single Assessment Numeric Evaluation (SANE), and the Veteran Rand 12-Item and 12-Item Short Form Health Survey (VR/SF12)] will be automatically emailed to patients using an electronic platform (OBERD). Rate at which these forms are completed (compliance rate) before surgery, as well 1-year post surgery will be monitored through OBERD.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Verma, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Carla M. Edwards, Evanston, Illinois, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03653455/Prot_SAP_000.pdf